CLINICAL TRIAL: NCT07019727
Title: Anterior Cruciate Ligament Injury Prevention Program ESSKA/ESMA: A Comprehensive Approach to Reducing the Incidence of Knee Joint Injuries in Czech Sport
Brief Title: ESSKA/ESMA ACL Injury Prevention Program in Czech Sport
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk University (Other)
Collaborators: Brno University Hospital (Other); St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0944/2025
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-06

CONDITIONS: Double Leg Vertical Jump (DLVJ); Single Leg Squat (SLS); Single Leg Drop Landing (SLDL); Drop Jump Test (DJ Test)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants of the program will attend a workshop led by a trained physiotherapist or strength and conditioning coach, conducted under medical supervision. Based on the ESSKA/ESMA methodology 'ACL Prevention for All', a total of 12 five-minute exercise units will be included.
  Interventions: Procedure: ESSKA/ESMA 'ACL Prevention for All' methodology
- Control Group (No Intervention): The control group will consist of a total of 50 individuals from selected sports in which the prevention program will not be implemented. Testing in this group will take place at the same time as in the athletes undergoing the program, with a follow-up test conducted after four months.

INTERVENTIONS:
Procedure: ESSKA/ESMA 'ACL Prevention for All' methodology — A workshop led by a trained physiotherapist/strength and conditioning coach and conducted under medical supervision. Based on the ESSKA/ESMA 'ACL Prevention for All' methodology, a total of 12 exercise units lasting 5 minutes each will be included.
  Arms: Intervention Group

SUMMARY:
This study aims to address the rising incidence of ACL injuries, particularly among adolescents, by developing and implementing a comprehensive prevention program based on the evidence-based "ACL Prevention for ALL" framework recommended by ESSKA-ESMA. The project focuses on muscle strengthening, flexibility, coordination, proper movement techniques, and a multidisciplinary approach involving coaches, physiotherapists, and physicians. Through targeted exercise modules, education, and dynamic evaluation-including 2D motion analysis-the study seeks to reduce ACL injuries, enhance movement safety, and enable individualized training plans by identifying and correcting muscle and biomechanical imbalances.

DETAILED DESCRIPTION:
1. Introduction According to published data, there has been a continuous increase in ACL (anterior cruciate ligament) injuries in developed countries over the last two decades. This trend has also been observed in the Czech Republic, based on analysis conducted by our expert group. The increase is particularly notable among adolescents. Knee joint injuries subsequently lead to reduced athletic performance and, in extreme cases, can prevent a return to competitive or elite-level sport. These injuries also have significant psychosocial consequences for young athletes.

   The evidence-based program "ACL Prevention for ALL," recommended by the professional society ESSKA-ESMA for widespread implementation, has been shown to reduce the incidence of ACL injuries by 50-60% across age groups and competitive levels. The prevention concept is based on several key components:

   Muscle Strengthening and Balance: Focusing on strengthening the thigh muscles (quadriceps and hamstrings) and ensuring their balance, which plays a critical role in knee stabilization.

   Flexibility: Improving lower limb flexibility can help reduce injury risk in individuals with reduced joint mobility.

   Coordination and Proprioceptive Training: Exercises that enhance coordination and body awareness improve athletes' ability to respond quickly to movement changes, reducing injury risk.

   Movement Technique: Teaching proper techniques for jumping, landing, and changing direction is essential to reduce mechanical stress on the knees.

   Multidisciplinary Approach: Involvement of coaches, physiotherapists, and physicians in the development and implementation of prevention programs tailored to athletes' specific needs.
2. Project Goals Reduce ACL Injury Incidence: Lower the occurrence of ACL injuries through targeted preventive exercise modules.

   Educate on Protective Movement Patterns: Teach jumping, landing, and change-of-direction techniques to minimize injury risk.

   Increase Awareness: Educate athletes, coaches, and healthcare professionals about injury risks and prevention strategies.

   Dynamic Evaluation: Regular monitoring and evaluation of program effectiveness to adapt and improve preventive measures based on current findings and results.

   The aim of the proposed research project is to develop and assess a methodology for identifying and correcting muscular imbalances and biomechanical deficiencies as part of a comprehensive ACL injury prevention program. The project will include an analysis of the effectiveness of various exercise and rehabilitation interventions, including 2D movement analysis, and their impact on muscular balance and technique. Final results and statistical data analysis will allow individualized training plans for athletes.
3. Methodology Initial Biomechanical Assessment

   Description: Lower limb landing biomechanics will be measured using Dartfish Express (2D analysis) at the start.

   Criteria Assessed:

   Double Leg Vertical Jump (DLVJ)

   Single Leg Squat (SLS)

   Single Leg Drop Landing (SLDL)

   Drop Jump Test (DJ Test)

   Workshop Implementation

   Description: Program participants will attend a workshop led by a trained physiotherapist/conditioning coach under medical supervision. Following ESSKA/ESMA's "ACL Prevention for ALL" methodology, 12 sessions of 10 minutes each will be conducted.

   Follow-up Measurement (3 Months)

   Description: After approximately 2,000 repetitions of correct movement execution, a follow-up 2D movement analysis will be conducted.

   Evaluation: Movement analysis results will be compared to assess the program's effectiveness in pilot sports.

   Pilot Sport Selection

   Description: Based on available data, five sports with the highest ACL injury incidence will be selected for the pilot.

   Sports: Football, basketball, volleyball, handball, floorball

   Participants: 10 males and 10 females per sport

   Statistical Analysis

   Description: Collected data will be analyzed using statistical methods, including ANOVA, to assess significance.

   Six-Month Follow-up

   Description: A second follow-up after six months will assess the sustainability of preventive effects and the occurrence of new injuries.

   Control Group Comparison

   Description: A control group of 50 individuals from the selected sports will not undergo the preventive program and will be tested at the same intervals.

   Evaluation: Results will be compared to those of the intervention group to verify program effectiveness.

   This structured methodological approach enables a comprehensive evaluation of the prevention program's effectiveness, supporting project goals and improving athlete health and performance.
4. Expected Outcomes Improved Muscle Balance and Strength: Increased balance between antagonistic muscle groups (e.g., quadriceps and hamstrings), documented via regular 2D biomechanical analyses.

   Long-term Performance Enhancement: Reduced injuries and improved biomechanics are expected to enhance overall athletic performance, measured through performance tests.

   More Effective Training Programs: Development and validation of effective and easily implementable training and rehabilitation programs, adjusted based on feedback and results.

   Increased Awareness and Knowledge: Raised awareness among athletes, coaches, and sports federation medical committees about injury risks and prevention strategies, supported by collected data.

   Reduced ACL Injury Incidence: Preventive program implementation is expected to significantly reduce ACL injury incidence in the target athlete group.

   Lower Injury Treatment Costs: Expected reduction in healthcare and rehabilitation costs due to fewer injuries.

   ACL Injury Registry and Monitoring: Establishment of a national ACL injury registry under the Czech Olympic Committee and sports federations, improving epidemiological data for program monitoring.
5. Implementation of Results in Practice Development of Standardized Training Programs / Integration of ESSKA/ESMA Program into Routine Training

   Develop standardized training programs based on research findings that include specific exercises to enhance muscle strength, balance, and movement technique.

   Include proven preventive techniques that reduce ACL injury incidence.

   Training for Coaches and Professionals

   Organize workshops and training sessions for coaches, physiotherapists, and other sports medicine professionals to familiarize them with new methodologies and targeted training approaches.

   Provide educational materials that incorporate the latest research and recommended injury prevention practices.

   Individual Athlete Assessment

   Implement regular assessments using methods such as 2D movement analysis to identify muscular imbalances and biomechanical deficiencies.

   For athletes identified with potential risks (P4 and P5), refer to gait laboratories for 3D motion analysis.

   Customize training programs to individual athletes' needs based on assessment results.

   Education and Awareness

   Create informational materials for athletes, coaches, and sports federation medical committees on injury prevention and the importance of muscle balance and movement technique.

   Disseminate validated information through seminars, online courses, social media, or publications.

   Publish results in peer-reviewed journals and foster international collaboration with IOC and ESSKA/ESMA.
6. Conclusion The primary objective and outcome of this project is to reduce ACL injury incidence in elite sports. A secondary objective is the protection of other knee joint structures that are frequently injured in conjunction with the ACL. Another crucial factor is the education of coaches, athletes, and healthcare personnel in prevention and proper movement techniques. Interdisciplinary collaboration-between sports medicine, physiotherapy, and coaching-is essential for effective implementation of the preventive approach.

Implemented recommendations and exercise protocols must be continuously updated based on the latest scientific evidence and practical experience. Long-term monitoring and evaluation of program effectiveness are key to ensuring success and sustainability. Based on international data, it is already evident that integrating the program into daily sports training is highly effective. The clear methodology and standardized evaluation format make it easy to implement the prevention program across all sports and age categories.

ELIGIBILITY:
Inclusion Criteria:

* Age group: Participants aged 17-20 years

Sports activity: Individuals actively engaged in sports with a high risk of ACL injury

Health status: Participants with no or minimal previous knee joint injuries that do not limit their current physical activity

Willingness to participate: Agreement to take part in the prevention program, including regular training and assessments

Informed consent: Signed informed consent for participation in the program and testing procedures; for minors, consent must be signed by legal guardians

Exclusion Criteria:

Current injury: Individuals with a current knee joint injury requiring treatment or surgery

Chronic conditions: Participants with chronic diseases or conditions that may affect the outcome of injury prevention (e.g., congenital abnormalities, neuromuscular disorders, or cardiovascular diseases)

Insufficient consent: Individuals who are unable or unwilling to provide written informed consent

Irregular participation: Individuals who do not comply with regular participation in the training program or assessments

Ages: 17 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak knee abduction moment | 4 months
  The strongest predictor of ACL injury risk according to the 'ligament dominance theory' and also the most frequently reported as changed after an IPP (Injury Prevention Program). Advantage: Quantifiable, measurable using 3D analysis and force platforms, and sensitive to changes.
Peak knee flexion angle | 4 months
  According to the 'quadriceps dominance theory,' a low angle increases the risk of ACL injury. Meta-analyses show an increase in the angle after IPP.
  Advantage: Easily measurable and consistently monitored in the literature.
Dynamic knee valgus (DKV) | 4 months
  Dynamic valgus is often described as a key injury mechanism, although its measurement is more complex and less standardized. It can be supplemented with specific angles such as knee abduction angle at initial contact (IC) and medial knee displacement.

SECONDARY OUTCOMES:
Peak hip flexion angle & hip flexion at initial contact | 4 months
  Lower flexion means higher vertical ground reaction force (vGRF) and lower force absorption, resulting in higher ACL load.
Vertical Ground Reaction Force (vGRF) | 4 months
  Higher vGRF at landing correlates with increased knee loading. The effect of IPP here is debatable, but it is relevant as a secondary parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Masaryk University, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol